CLINICAL TRIAL: NCT03465163
Title: Safety and Efficacy of a Deep Brain Stimulation System in Epilepsy: A Feasibility Study for Tracking Neural Excitability
Brief Title: A Deep Brain Stimulation System in Epilepsy: Tracking Neural Excitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Mark Cook, Principal Investigator, St Vincent's Hospital Melbourne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HREC/17/SVHM/146
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Epilepsy; Nodular Heterotopia
MeSH Terms: conditions — Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Recovery (No Intervention): Two months recovery (no stimulation) following bilateral implantation of Medtronic PC+S devices into the anterior nucleus of the thalamus and the hippocampus. Thirty second EEG snapshots will be recorded every 15 minutes
- Baseline (No Intervention): No stimulation, 30 second EEG snapshots recorded every 15 minutes We require a minimum of 5 seizures to occur during this phase.
- Probing (Experimental): Deep Brain Stimulation Electrically stimulate the thalamus continuously at a low frequency (2Hz). Thirty second EEG snapshots recorded every 15 minutes.
  We require a minimum of 5 seizures to occur during this phase.
  Interventions: Device: Deep Brain Stimulation
- Probe Calibrated Deep Brain Stimulation (Experimental): Deep Brain Stimulation In this phase we explore 18 deep brain stimulation parameter configurations (three stimulus intensities; 3,4,5 Volts, six different frequencies; 125 130, 135, 140,145, 150 Hz) during two of the clinic visits. Each deep brain stimulation parameter configuration will be tested for 1 minute with 4 minutes between each configuration test. The probing responses will be used to optimise the deep brain stimulation parameters for each participant. This phase of the study continues for 2 months.
  Interventions: Device: Deep Brain Stimulation
- Open Deep Brain Stimulation (Experimental): Deep Brain Stimulation During this phase the deep brain stimulation parameters may be altered from the probing optimised parameters according to patient needs.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — The device is called the Medtronic Activa PC+S system. Two devices will be implanted per participant. The electrodes will be surgically implanted bilaterally into the hippocampus and anterior nucleus of the thalamus.
  Other Names: DBS
  Arms: Open Deep Brain Stimulation; Probe Calibrated Deep Brain Stimulation; Probing

SUMMARY:
The main purpose of this research project is to evaluate the safety and effectiveness of a surgically implanted device called the Medtronic Activa PC+S System in patients with medically refractory epilepsy (people who have seizures that are not completely controlled by medical therapy). The system sends small electrical pulses into a part of the brain called the thalamus to help control seizures. It sends this signal in regularly, regardless of if a seizure is occurring. A different version of this device is already approved for the treatment of epilepsy in Australia. This study aims to use the brain's responses to single pulse electrical stimulation to measure the level of seizure susceptibility. The investigators would like to show that this measure can be used to provide more effective deep brain stimulation therapies, to stop seizures.

ELIGIBILITY:
Inclusion Criteria:

Patients with epilepsy with non-resectable pathologies, or clearly defined focal seizures without a defined structural pathology.

Patients will be required to have a seizure diary (of up to 3 months) recording at least five seizures per month that are well separated in time (at least 8 hours apart).

Exclusion Criteria:

Previous diagnosis of psychogenic/non-epileptic seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Seizure Rate | Recorded throughout the baseline (2-4 months post implant) and probe calibrated DBS phase( 6-8 months post implant)
  Comparing the number of seizures per patient, as recorded by Medtronic Activa PC+S system in the baseline vs. probe calibrated DBS phase.

SECONDARY OUTCOMES:
Determine if probing responses provide a seizure susceptibility measure. | Throughout probing phase (4-6 months post implant)
  Calculate probability of seizure in the near future given the features of the probing response shape during pre-ictal and inter-ictal periods on training dataset and then test predictive power on remaining data. Features defining the probing response shape will include peak amplitude and peak latency. Seizure occurrences will be determined by the Medtronic PC+S device.
Change in brain excitability following DBS treatment, assessed according to changes in probing response energy before and after stimulation therapy. | Throughout probing phase (4-6 months post implant) and probe calibrated DBS phase (6-8 months post implant).

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital Melbourne, Melbourne, Victora, Australia

IPD SHARING:
Plan to Share IPD: No